CLINICAL TRIAL: NCT03256084
Title: Characterization of Tumoral Circulating Cells According to Stage of Progression of Colorectal Cancers
Brief Title: Tumoral Circulating Cells and Colorectal Cancer Progression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut Paoli-Calmettes (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Beckman Coulter, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CTC-Côlon-IPC 2015-020
Record Dates: First submitted 2017-06-19; First posted 2017-08-21 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Colorectal Cancer (Experimental): Localized stage II/III (group 1), metastatic non resectable (group 2), metastatic potentially resectable (group 3).
  Additional blood samples specific for the research will be collected. Tissue samples will be taken on surgical specimens from surgery.
  Interventions: Procedure: Blood and tumor samples

INTERVENTIONS:
Procedure: Blood and tumor samples — Blood and tumor samples

SUMMARY:
Prospective research of circulating tumor cells as markers of progression risk in colorectal cancer.

DETAILED DESCRIPTION:
This study aims at allowing a better understanding of which circulating tumor cells (CTC) have the higher risk of metastasis of in the overall population of CTC.

Prospective monocenter open-label study.

In the frame of the management of the disease, blood samples will be collected at different times of treatment, regarding disease status (localized of stage II/III, metastatic non resectable, metastatic potentially resectable). Tissue samples will be collected for patients scheduled for surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patient of more than 18 years old
2. Histological diagnosis of colic adenocarcinoma metastatic or not
3. Before any treatment with systemic chemotherapy
4. Patient affiliated to, or beneficiating of the national security
5. Patient having signed informed consent

Exclusion Criteria:

1. Patient with previous chemothrapy treatment
2. Patient with more than one evolutive tumoral pathology
3. Patient under long-term immunosuppressor treatment
4. Patient with severe infection
5. Pregnant or breasting woman
6. Person in an emergency situation, adult subject to a legal protection measure (a guardian, guardianship or safeguard of justice), or unable of expressing his / her consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-07-17 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Evaluation of CTC features | Group 1: at surgery, 4 (+/- 1) weeks post-surgery, at progression. Group 2: before chemotherapy, after 4 months treatment (responders), at progression. Group 3: before neoadjuvant surgery, at surgery, 4 (+/- 1) weeks post-surgery, at progression.
  Changes in the number of CTC with high risk to form metastasis, defined as an aggregation of phenotypic, molecular and functional characteristics.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc RAOUL, Pr, Study Director — Institut Paoli-Calmettes
Locations (1):
- Institut Paoli Calmettes, Marseille, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sotelo MJ, Sastre J, Maestro ML, Veganzones S, Vieitez JM, Alonso V, Gravalos C, Escudero P, Vera R, Aranda E, Garcia-Alfonso P, Gallego-Plazas J, Lopez C, Pericay C, Arrivi A, Vicente P, Ballesteros P, Elez E, Lopez-Ladron A, Diaz-Rubio E. Role of circulating tumor cells as prognostic marker in resected stage III colorectal cancer. Ann Oncol. 2015 Mar;26(3):535-41. doi: 10.1093/annonc/mdu568. Epub 2014 Dec 15. PMID 25515656
- [Result] Hodgkinson CL, Morrow CJ, Li Y, Metcalf RL, Rothwell DG, Trapani F, Polanski R, Burt DJ, Simpson KL, Morris K, Pepper SD, Nonaka D, Greystoke A, Kelly P, Bola B, Krebs MG, Antonello J, Ayub M, Faulkner S, Priest L, Carter L, Tate C, Miller CJ, Blackhall F, Brady G, Dive C. Tumorigenicity and genetic profiling of circulating tumor cells in small-cell lung cancer. Nat Med. 2014 Aug;20(8):897-903. doi: 10.1038/nm.3600. Epub 2014 Jun 1. PMID 24880617
- [Result] Yu M, Bardia A, Aceto N, Bersani F, Madden MW, Donaldson MC, Desai R, Zhu H, Comaills V, Zheng Z, Wittner BS, Stojanov P, Brachtel E, Sgroi D, Kapur R, Shioda T, Ting DT, Ramaswamy S, Getz G, Iafrate AJ, Benes C, Toner M, Maheswaran S, Haber DA. Cancer therapy. Ex vivo culture of circulating breast tumor cells for individualized testing of drug susceptibility. Science. 2014 Jul 11;345(6193):216-20. doi: 10.1126/science.1253533. PMID 25013076
- [Result] Khoo BL, Lee SC, Kumar P, Tan TZ, Warkiani ME, Ow SG, Nandi S, Lim CT, Thiery JP. Short-term expansion of breast circulating cancer cells predicts response to anti-cancer therapy. Oncotarget. 2015 Jun 20;6(17):15578-93. doi: 10.18632/oncotarget.3903. PMID 26008969
- See also: Official Website of the Sponsor — http://institutpaolicalmettes.fr